CLINICAL TRIAL: NCT01121666
Title: A Phase III Assessor-blinded Randomized Parallel Group Multi-centre Study to Compare Efficacy and Safety of Two r-hFSH Formulations (AFOLIA Versus Gonal-f) in Women for Assisted Reproductive Treatment
Brief Title: Multi-centre Study to Compare Efficacy and Safety of AFOLIA and Gonal-f in Women for Assisted Reproductive Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Finox AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIN3001; 2010-019287-37 (EudraCT Number)
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Infertility
Keywords: Assisted reproductive treatment; Superovulation; Follitropin alfa; r-hFSH; AFOLIA
MeSH Terms: conditions — Infertility | interventions — follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gonal-f® (Follitropin alfa) (Active Comparator)
  Interventions: Drug: Follitropin alfa
- AFOLIA-150 (Follitropin alfa) (Experimental)
  Interventions: Drug: Follitropin alfa

INTERVENTIONS:
Drug: Follitropin alfa — 150IU per day subcutaneously for a maximum of 16 days

SUMMARY:
Ther purpose of this study is to show equivalence between AFOLIA and Gonal-f® with regard to the number of oocytes retrieved in women for assisted reproductive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 38 years with regular menstrual cycles of 25-35 days
* First or second cycle in the present series of ART
* BMI ≥ 18 ≤ 30 kg/m2
* Basal FSH < 10 IU/L (cycle day 2-5)
* E2 levels < 50pg/mL (< 0.18 nmol/L) at the day of FSH administration
* Antral follicle count (AFC) ≥ 10 to ≤ 25 follicles (sum of both ovaries)
* Infertility due to any of the following factors: tubal factor, mild endometriosis (ASRM stage 1-2), male factor, unexplained infertility
* Presence of both ovaries and normal uterine cavity (confirmed by transvaginal ultrasound within 6 months before randomisation)
* Willingness to participate in the study and to comply with the study protocol
* Informed consent

Exclusion Criteria:

* Presence of pregnancy
* History of ≥2 succeeding ART cycles (IVF and/or ICSI) before the study cycle without clinical pregnancy
* Presence of clinically significant systemic disease
* Presence of chronic cardiovascular, hepatic, renal or pulmonary disease
* Presence of uncontrolled endocrine disorder
* Previous history or presence of severe ovarian hyperstimulation syndrome
* Presence of polycystic ovaries (PCO)
* Presence of severe endometriosis (ASRM stage 3 or stage 4) and hydrosalpinx
* Neoplasia, including tumors of the hypothalamus and pituitary gland
* Abnormal bleeding of undetermined origin
* History of poor response to gonadotropin treatment (defined as fewer than 5 oocytes retrieved in a previous attempt)
* Male infertility without mobile spermatozoa in the ejaculate, that need testicular of epididymal sperm retrieval (MESA/TESE/TESA)
* Endocrine abnormality such as TSH or prolactin level elevations outside the reference range if clinically relevant at screening
* Any hormonal treatment within 1 month before the start of the FSH treatment (with the exception of levothyroxin)
* History of drug, nicotine or alcohol abuse within the last 12 months (> 10 cigarettes/day)
* Administration of other investigational products within the last month
* Clinically abnormal findings at Visit 1
* Planned PGS/PGD/PBB or assisted hatching
* Concomitant participation in an other study protocol
* History of extrauterine pregnancy in the previous 3 months
* Known allergy or hypersensitivity to progesterone or to any of the excipients (including peanut oil) of the additional study medication (GnRH agonist, vitrelle®, and Utrogestan®)
* Presence or history of thrombophlebitis or thromboembolic disorders
* Presence or history of cerebral haemorrhage
* Presence or history of porphyria

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 460 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Imthurn, Principal Investigator — University of Zurich
Locations (16):
- Austria (5):
  - Kinderwunsch Institut Schenk GmbH, Graz
  - Landes-Frauenklinik und Kinderklinik Linz, Linz
  - AKH Vienna, Vienna
  - IVF Zentrum Döbling, Vienna
  - Privatspital Goldenes Kreuz, Vienna
- Denmark (3):
  - Fertility Clinic, Copenhagen
  - Copenhagen Fertility Center, Copenhagen
  - Dansk Fertilitetsklinik, Frederiksberg
- Germany (2):
  - Universitätsklinikum Bonn, Bonn
  - Universitäts-Frauenklinik, Heidelberg
- Spain (2):
  - Institut Universitari Dexeus, Barcelona
  - IVI Madrid, Madrid
- University Hospital of Zurich, Zurich, Switzerland
- United Kingdom (3):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Kings College Hospital, London
  - St Barthlomew's Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 15 centers in six European countries from July 2010 until April 2012.
Pre-assignment Details: Of 460 participants in this trial 88 were reported as screening failures prior the group assignment.
Period: Overall Study
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Started | 249 | 123
Completed | 220 | 113
Not Completed | 29 | 10
Not completed — Protocol Violation | 29 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa) | Total
Number analyzed (Participants) | 249 | 123 | 372
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (4.02) | 32.1 (3.76) | 31.95 (3.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249 | 123 | 372
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 229 | 117 | 346
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  Austria | 88 | 43 | 131
  Denmark | 75 | 37 | 112
  Spain | 33 | 19 | 52
  Germany | 24 | 11 | 35
  United Kingdom | 21 | 10 | 31
  Switzerland | 8 | 3 | 11
FSH baseline concentration [Mean (Full Range); unit: (IU/L)] — The FSH concentration was measured at baseline in IU/L.
  (IU/L) | 6.9 [2.5 to 17.1] | 6.9 [2.8 to 10] | 6.9 [2.5 to 17.1]
Antral follicle count [Mean (Full Range); unit: Antral follicle count] | 15.1 [10 to 24] | 15.3 [10 to 24] | 15.2 [10 to 24]
Body Mass Index [Mean (Full Range); unit: kilogramm/ square meter] | 22.7 [18.0 to 30.3] | 22.4 [18.2 to 28.7] | 22.6 [18.0 to 30.3]
GnRH-agonist duration [Mean (Full Range); unit: days] | 23.5 [11.0 to 44.0] | 22.7 [12.0 to 46.0] | 23.1 [11.0 to 46.0]
AMH less than 24 pmol/L [Number; unit: Number of participants] — Number of patients of each group who had a lower AMH level than 24 pmol/L. The cut-off level was defined on the basis of the evaluated level published previously.
  Number of participants | 106 | 47 | 153

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved (Per Protocol Population)
Description: As soon as ovulation criteria were reached, HCG was given to trigger ovulation and 34-36 hours later, oocytes were retrieved. If criteria for ovulation triggering could not be reached by FSH stimulation on day 16, treatment was to be stopped.
  The equivalence in the number of retrieved oocytes was tested using a pre-determined clinical equivalence margin of +/- 2.9 oocytes
Time Frame: 34-36 hours after hCG administration and after maximum 16 days of r-hFSH treatment
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: Number of retrieved oocytes
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 220 | 113
Number of retrieved oocytes | 10.8 (5.11) | 10.6 (6.06)
Statistical Analysis 1: Comparison: AFOLIA-150 (Follitropin Alfa) vs Gonal-f® (Follitropin Alfa); This study was powered to test equivalence using a two one-sided test (TOST) of the number of oocytes retrieved; Test type: Non-Inferiority or Equivalence — This study was powered to test equivalence using a two one-sided test (TOST) of the number of oocytes retrieved with a power of 90%, an alpha error of 2.5% and a pre-determined clinical equivalence margin of +/-2.9 oocytes for the relevant population; p = 0.0003, Shuirmann's TOST — This study was powered to test equivalence using a two one-sided test (TOST) with a power of 90%, an alpha error of 2.5% and a pre-determined clinical equivalence margin of +/-2.9 oocytes for the relevant population

2. Secondary Outcome: Number and Size of Follicles ≥ 12 mm at Day 8 of Stimulation
Description: The number and size of follicles 12 mm or over in diameter at day 8 of stimulation were evaluated as secondary end-point.
Time Frame: Day 8 of stimulation
Population: All participants were analyzed.
Measure: Mean (Standard Deviation); unit: Number of follicles
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Number of follicles
  ≥ 12 mm | 11.8 (4.73) | 11.1 (4.23)
  ≥ 15 mm | 8.3 (3.81) | 7.7 (3.60)
  ≥ 17 mm | 4.9 (3.29) | 4.5 (2.71)
Statistical Analysis 1: Comparison: AFOLIA-150 (Follitropin Alfa) vs Gonal-f® (Follitropin Alfa); Test type: Superiority or Other; p = 0.2357, Wilcoxon (Mann-Whitney) — Follicles of 12 mm
Statistical Analysis 2: Comparison: AFOLIA-150 (Follitropin Alfa) vs Gonal-f® (Follitropin Alfa); Test type: Superiority or Other; p = 0.1395, Wilcoxon (Mann-Whitney) — Follicles of 15 mm
Statistical Analysis 3: Comparison: AFOLIA-150 (Follitropin Alfa) vs Gonal-f® (Follitropin Alfa); Test type: Superiority or Other; p = 0.3992, Wilcoxon (Mann-Whitney) — Follicles of 17 mm

3. Secondary Outcome: E2 Concentration at Day 8 and at Day of hCG Administration
Description: The serum concentration of oestradiol was assessed at day 8 and the day of hCG administration.
Time Frame: Day 8 of stimulation and at the day of hCG administration (after max. 16 days of r-FSH treatment)
Population: All participants were analyzed.
Measure: Mean (Standard Deviation); unit: pmol/ L
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
pmol/ L
  Day of hCG administration | 8982.3 (6535.3) | 7704.2 (5345.8)
  Day 8 | 3958.9 (3699.4) | 3234.0 (2428.1)

4. Secondary Outcome: Total Dose of r-hFSH Administered
Description: Total dose of r-hFSH required was assessed.
Time Frame: Day of hCG administration (after maximum 16 days of r-hFSH treatment)
Population: All participants were analyzed.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
IU | 1555.7 (293.00) | 1569.2 (259.20)
Statistical Analysis 1: Comparison: AFOLIA-150 (Follitropin Alfa) vs Gonal-f® (Follitropin Alfa); Test type: Superiority or Other; p = 0.9638, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Quality of Oocytes Retrieved
Description: Number of patients with ovum pick-up
Time Frame: 34-36 hours after hCG administration
Population: Intention to treat population
Measure: Number; unit: Participants
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Participants
  day 2 | 82 | 36
  day 3 | 53 | 28

6. Secondary Outcome: Fertilisation Rate of Oocytes
Description: Fertilisation rate was assessed
Time Frame: 1 day after ovum pick-up
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: percentage of oocytes
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
percentage of oocytes | 66.1 (24.84) | 64.0 (24.76)

7. Secondary Outcome: Embryo Quality: Mean Number of Blastomeres
Description: Main embryo quality parameter "mean number of blastomeres"
Time Frame: Day 2 of OPU/fertilisation
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: Number of blastomeres at day 3
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Number of blastomeres at day 3 | 6.6 (2.41) | 6.4 (2.49)

8. Secondary Outcome: Number of Participants With Cryopreserved 2PNs, Embryos/Blastocysts
Time Frame: Day 1, 2, 3 and 5 of OPU/fertilisation
Population: Intention to treat population
Measure: Number; unit: Patients with cryopreservation
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Patients with cryopreservation | 103 | 55

9. Secondary Outcome: Number of Days of r-hFSH Stimulation
Description: Mean duration of stimulation was assessed.
Time Frame: At the day of hCG administration, up to 16 days
Population: All participants were analyzed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
days | 10.6 (1.91) | 10.7 (1.72)
Statistical Analysis 1: Comparison: AFOLIA-150 (Follitropin Alfa) vs Gonal-f® (Follitropin Alfa); Test type: Superiority or Other; p = 0.8926, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Number of Patients With Cycle Cancellation
Description: Number of patients with cycle cancellation was assessed.
Time Frame: Until child birth/miscarriage, up to the end of the study
Population: Intention to treat population
Measure: Number; unit: Number of patients
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Number of patients | 13 | 5

11. Secondary Outcome: Number of Patients With Good Response
Description: Good response was defined as "patients with an oocyte retrieval of four or more oocytes"
Time Frame: Until child birth/miscarriage, up to the end of the study
Population: Intention to treat population.
Measure: Number; unit: Participants
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Participants | 217 | 107

12. Secondary Outcome: Implantation Rate
Description: Defined as fetal sac per embryo transferred.
Time Frame: Five to six weeks after oocyte retrieval
Population: Intention to treat population.
Measure: Number; unit: Percentage of implantations
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Percentage of implantations | 31.8 | 36.7

13. Secondary Outcome: Clinical Pregnancy Rate
Description: Presence of at least one intrauterine gestational sac.
Time Frame: Five to six weeks after oocyte retrieval
Population: Intention to treat population
Measure: Number; unit: Clinical pregnancies
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Clinical pregnancies | 90 | 55

14. Secondary Outcome: Ongoing Pregnancy
Description: Ongoing pregnancy per embryo transfer. Presence of at least one viable fetus 10 weeks after embryo transfer.
Time Frame: Ten weeks after embryo transfer
Population: Intention to treat population
Measure: Number; unit: Ongoing pregnancies
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Ongoing pregnancies | 84 | 51

15. Secondary Outcome: Live Birth Rate
Description: Patients with liveborn children
Time Frame: After childbirth with questionnaire
Population: Intention to treat population
Measure: Number; unit: Patients with liveborn children
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Patients with liveborn children | 80 | 51

16. Primary Outcome: Number of Oocytes Retrieved (Intention-to-treat Population)
Description: as for outcome 1
Time Frame: 34-36 hours after hCG administration and after maximum 16 days of r-hFSH treatment
Population: Intention-to-treat population
Measure: Mean (Standard Deviation); unit: Number of retrieved oocytes
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Number of retrieved oocytes | 10.7 (5.62) | 10.4 (6.14)
Statistical Analysis 1: Comparison: AFOLIA-150 (Follitropin Alfa) vs Gonal-f® (Follitropin Alfa); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0003, Shuirmann's TOST

17. Secondary Outcome: Embryo Quality: Absence of Multinucleation
Description: Main embryo quality parameter "absence of multinucleation" observed.
Time Frame: Day 3
Population: Intention to treat population
Measure: Number; unit: Percentage of absent multinucleation
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Percentage of absent multinucleation | 93.6 | 93.9

18. Secondary Outcome: Quality of Oocytes Retrieved
Description: Number of patients with transferred blastocysts
Time Frame: At day 4 and 5
Population: Intention to treat population
Measure: Number; unit: Participants
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Participants
  day 4 | 10 | 2
  day 5 | 76 | 46

19. Secondary Outcome: Quality of Oocytes Retrieved
Description: Number of embryos per blastocysts transferred
Time Frame: Day of embryo transfer, either 2, 3 or 5 days after oocyte retrieval
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: embryos per blastocysts transferred
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
embryos per blastocysts transferred | 1.5 (0.52) | 1.6 (0.53)

20. Secondary Outcome: Clinical Pregnancy Rate (Second Treatment Cycle)
Description: Presence of at least one intrauterine gestational sac.
Time Frame: Five to six weeks after oocyte retrieval
Population: Population with a second treatment cycle
Measure: Number; unit: Clinical pregnancies
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 72 | 38
Clinical pregnancies | 25 | 10

21. Secondary Outcome: Ongoing Pregnancy (Second Treatment Cycle)
Description: Ongoing pregnancy per embryo transfer. Presence of at least one viable fetus 10 weeks after embryo transfer.
Time Frame: 10 weeks after embryo transfer
Population: Population with a second treatment cycle
Measure: Number; unit: Ongoing pregnancies
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 72 | 38
Ongoing pregnancies | 22 | 9

22. Secondary Outcome: Quality of Oocytes Retrieved
Description: The maturity of the cumulus oophorus was assessed.
Time Frame: After oocyte retrieval, 34 to 36 hours after hCG administration
Population: Intention to treat population
Measure: Number; unit: Percentage of cumulus oophori
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Percentage of cumulus oophori
  very mature | 9.1 | 9.4
  mature | 75.7 | 75.3
  immature | 14.5 | 14.2

23. Secondary Outcome: Quality of Oocytes Retrieved
Description: The nuclear maturity was assessed (Germinal vesicle, Metaphase I, Metaphase II).
Time Frame: After oocyte retrieval, 34 to 36 hours after hCG administration
Population: Intention to treat population
Measure: Number; unit: Percentage of cells
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Number analyzed (Participants) | 249 | 123
Percentage of cells
  Germinal vesicle | 9.5 | 9.1
  Metaphase I | 7.2 | 7.7
  Metaphase II | 83.4 | 83.3

ADVERSE EVENTS:
Time Frame: Study period + 30 days
Arm/Group | AFOLIA-150 (Follitropin Alfa) | Gonal-f® (Follitropin Alfa)
Serious Adverse Events (participants affected / at risk) | 12/249 | 3/123
Other Adverse Events (participants affected / at risk) | 182/249 | 83/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AFOLIA-150 (Follitropin Alfa) (N=249) | Gonal-f® (Follitropin Alfa) (N=123)
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Ovarian haemorrhage (Reproductive system and breast disorders) | 1 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 7 | 2
Syncope (Nervous system disorders) | 0 | 1
Body temparature increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AFOLIA-150 (Follitropin Alfa) (N=249) | Gonal-f® (Follitropin Alfa) (N=123)
Injection site erythema (General disorders) | 68 | 44
Injection site haematoma (General disorders) | 60 | 19
Headache (Nervous system disorders) | 55 | 25
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 55 | 16
Injection site pain (General disorders) | 39 | 21
Nausea (Gastrointestinal disorders) | 23 | 6
Injection site swelling (General disorders) | 15 | 10
Abdominal distension (Gastrointestinal disorders) | 14 | 6
Fatigue (General disorders) | 13 | 4
Abdominal pain (Gastrointestinal disorders) | 13 | 6
Abdominal pain upper (Gastrointestinal disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No